CLINICAL TRIAL: NCT02134964
Title: A Phase 1, Randomized, Dose Escalation, Single Center, Safety and Pharmacokinetic Study of Single and Multi-Dose, Orally Administered OLT1177 Capsules in Healthy Subjects
Brief Title: Phase 1 Safety and PK Study of OLT1177 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OLT1177-04
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Pharmacokinetics; Dose escalation; Randomized; Healthy volunteers; OLT1177; Olatec
MeSH Terms: interventions — dapansutrile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- OLT1177 Capsules (Experimental): A total of 5 patients in each cohort will receive OLT1177 Capsules:
  * Cohort 1 will receive a single 100 mg dose of OLT1177
  * Cohort 2 will receive a single 300 mg dose of OLT1177
  * Cohort 3 will receive two 1000 mg doses of OLT1177 (seven days apart)
  * Cohort 4 will receive 100 mg doses of OLT1177 QD for 8 days
  * Cohort 5 will receive 300 mg doses of OLT1177 QD for 8 days
  * Cohort 6 will receive 1000 mg doses of OLT1177 QD for 8 days
  Interventions: Drug: OLT1177 Capsules
- Placebo Capsules (Placebo Comparator): A total of 1 patient in each cohort will receive Placebo Capsules:
  * Cohort 1 will receive a single placebo capsule
  * Cohort 2 will receive three placebo capsules
  * Cohort 3 will receive ten placebo capsules (seven days apart)
  * Cohort 4 will receive a single placebo capsule QD for 8 days
  * Cohort 5 will receive three placebo capsules QD for 8 days
  * Cohort 6 will receive ten placebo capsules QD for 8 days
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: OLT1177 Capsules — OLT1177 Capsules are an experimental drug.
  Arms: OLT1177 Capsules
Drug: Placebo Capsules — Placebo Capsules are identical in all ways to the study drug, but contain no active pharmaceutical ingredient.
  Arms: Placebo Capsules

SUMMARY:
This study is a randomized, placebo-controlled, sequential ascending-dose study of healthy volunteers after administration of single or multiple dose(s) of investigational drug (OLT1177 Caps or Placebo Caps). A total of 36 subjects will be enrolled across 6 cohorts, and subjects in each cohort will be randomized in a ratio of 5 active to 1 placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years old, inclusive
* In good health as determined by the Investigator based on subject's medical history, ECG and physical examination at Baseline and safety laboratory tests (chemistry, hematology, coagulation and urinalysis) at Screening
* Normal blood pressure of 130/85 mmHg or lower
* Ability to provide written, informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the Investigator, to comply with all the requirements of the study

Exclusion Criteria:

* Women of childbearing potential, or men whose sexual partner(s) is a woman of childbearing potential who:

  1. Are or intend to become pregnant (including use of fertility drugs) during the study
  2. Are nursing
  3. Are not using an acceptable, highly effective method of contraception until all follow-up procedures are complete. (Acceptable, highly effective forms of contraception are defined as: oral contraception, intrauterine device, systemic [injectable or patch] contraception, double barrier methods, naturally or surgically sterile, strict abstinence or partner has been sterilized. If hormonal-based birth control is being used, subject or subject's sexual partner(s) must be on a stable-dose for ≥ 3 months prior to the Baseline visit and maintained at the same dosing level throughout the study.)
* Use of any drug treatment at the time of the study (with the exception of 81 mg aspirin and prescription oral or systemic contraceptives)
* Taking any prescription medications (other than oral or systemic contraceptives) within 14 days prior to administration of investigational drug or taking any over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 14 days prior to administration of investigational drug, except for topical products without systemic absorption
* Use of NSAIDs or other prescription pain medication, more than once or twice a week, especially if taken for chronic or frequently recurring headache
* Active infection within 3 days of the Baseline visit
* History of or known positive for HIV, Hepatitis B surface antigen (HBsAg) or antibodies to Hepatitis C Virus (HCV)
* Diagnosed with any form of internal cancer within the past 5 years
* Any other medical conditions, diseases or prior surgeries that in the opinion of the Investigator would impair the subject from safely participating in the trial and/or completing any protocol requirements
* History of anaphylactic reactions to any systemic or topical compounds
* Have donated plasma (500 mL) within 7 days prior to drug administration
* Have donated or lost whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows: 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration
* Is a user of any nicotine products (including chewing tobacco, snuff and/or e-cigarettes)
* Is not willing to restrict food or beverage including: alcohol, caffeine, poppy seeds, xanthine derivatives or xanthine-related compounds, energy drinks, natural health products, grapefruit juice, pomelo, Seville orange and marmalade use during the study as specified in Section 7.1.5
* Is lactose intolerant
* Is unable or unwilling to consume products containing bovine byproducts
* Is unable to adhere to or understand the requirements of the protocol
* If continuing on to Part B, subject is unable or unwilling to ingest the full study-provided high-fat breakfast within 30 minutes
* Enrollment in any trial and/or use of any Investigational Drug or device within the immediate 30-day period prior to the Baseline visit
* Enrollment in any study previously sponsored by Olatec Industries LLC, specifically Study OLT1177-01, Study OLT1177-02 or Study OLT1177-03

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Recording of adverse events | Screening through Day 28 follow-up
  Adverse events will be described with respect to seriousness, intensity, relationship to treatment, action taken and outcome of the event.

SECONDARY OUTCOMES:
Safety Laboratory Measurements | Screening through Day 15 (Part A&B)/Day 22 (Part C) visit
  Blood samples will be drawn and analyzed for: chemistry, hematology, lipids and coagulation.
Electrocardiogram | Screening through Day 15 (Part A&B)/Day 22 (Part C) visit
  Electrocardiograms will be captured and analyzed for changes throughout the duration of the study.
Vital Signs | Screening through Day 15 (Part A&B)/Day 22 (Part C) visit
  Vital signs (pulse, resting blood pressure, temperature and respirations) will be recorded and analyzed for changes throughout the duration of the study.
Physical Examination | Screening through Day 15 (Part A&B)/Day 22 (Part C) visit
  Physical examinations will be conducted to assess changes in subject health throughout the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Terry M Jones, MD, FAAD, Principal Investigator — J&S Studies
Locations (1):
- J&S Studies, Inc, College Station, Texas, United States